CLINICAL TRIAL: NCT03777553
Title: Narrative Exposure Therapy for Justice-Involved Veterans (D1298-W)
Brief Title: Narrative Exposure Therapy (NET)
Acronym: NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1298-W-1
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder; criminal justice; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a single group pre/post trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VETNET (Experimental): Narrative Exposure Therapy for Justice-Involved Veterans
  Interventions: Behavioral: Narrative Exposure Therapy for Justice-Involved Veterans

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy for Justice-Involved Veterans — Behavioral intervention that uses narrative therapy and exposure to address repeated or complex trauma.
  Other Names: VETNET

SUMMARY:
The purpose of this study is to learn more about Narrative Exposure Therapy for Justice Involved Veterans. This pilot study will examine the feasibility of this intervention in a justice-involved veteran population, and will see whether the intervention needs to be tailored to best meet their needs. The investigators will examine whether the intervention impacts key clinical outcomes, including posttraumatic stress disorder symptoms, as well as on measures of moral injury, anger, depression, suicidality, and aggression.

DETAILED DESCRIPTION:
The overall objective of this application is to gather data on the use of Narrative Exposure Therapy for Justice Involved Veterans (VETNET) in a pilot sample of justice-involved Veterans with PTSD, with a particular focus on obtaining data on feasibility and acceptability of the intervention in a justice-involved veteran population, and determining what further adaptations are needed to tailor this intervention to justice-involved Veterans (JIV). The investigators are also interested in evaluating whether the intervention has the potential to have an effect on key clinical outcomes, including posttraumatic stress disorder (PTSD) symptoms, as well as on measures of moral injury, anger, depression, suicidality, and aggression.

The following Specific Aims have been developed for this project:

Aim 1: Evaluate study feasibility and treatment delivery procedures of Narrative Exposure Therapy for Justice Involved Veterans (VETNET) in justice-involved Veterans (JIV) with PTSD. Data gathered will include recruitment rates, drop-out rates, adverse event frequency and severity, and participant engagement in treatment. As necessary, identify further adaptations that are needed to tailor this intervention specifically to JIV.

Aim 2: Evaluate the impact of VETNET on PTSD symptoms, as well as on related outcomes including moral injury, anger, depression, suicidality, and aggression.

ELIGIBILITY:
Inclusion Criteria:

* Is a veteran;
* Recent justice involvement including current probation, parole, or house arrest, or having been released from jail or prison within the past 1 year;
* Meets current criteria for PTSD.

Exclusion Criteria:

* Currently incarcerated;
* Current, active psychosis;
* Is at imminent risk for suicide or homicide warranting immediate intervention;
* Substance abuse that is severe enough to prevent full engagement in the study protocol;
* Concurrent trauma-focused psychotherapy including Prolonged Exposure Therapy, Cognitive Processing Therapy, or EMDR;
* Is unable to unwilling to complete study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Van Voorhees, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VETNET
Started | 9 (Participants who signed consent form and underwent screening.)
Completed | 5 (Participants who were eligible to participate, and who attended at least one NET session. All participants who attended at least one session completed the treatment protocol and the post-treatment measures. Four of the five completed the 3 months post-treatment measures.)
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Veterans with recent justice involvement including current probation, parole, or house arrest, or having been released from jail or prison within the past 1 year; and who met criteria for PTSD at the time of study entry.
Arm/Group | VETNET
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: PTSD Checklist for the DSM-5 (PCL-5)
Description: On the PCL-5 participants first report an autobiographical narrative of a trauma, and subsequently rate how bothered they were by each symptom (0 [not at all] - 4 [extremely]) for all DSM-V PTSD symptoms within the past week. Total score range is 0 to 80, with higher scores reflecting greater symptomatology. Positive change score reflects increase in PTSD symptoms from baseline to post-treatment; negative change score reflects decrease in PTSD symptoms from baseline to post-treatment.
Time Frame: Change in total score from baseline to end of treatment (approximately 10-12 weeks), and baseline to 3 months post-treatment.
Population: Veterans with recent justice involvement including current probation, parole, or house arrest, or having been released from jail or prison within the past 1 year, and who met criteria for posttraumatic stress disorder at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VETNET
Number analyzed (Participants) | 5
units on a scale
  baseline | 47.8 (15.0)
  post-treatment | 25.0 (18.6)
  3 months post treatment: number analyzed (Participants) | 4
  3 months post treatment | 20 (10.4)
  mean change score pre to post | -22.8 (9.0)
  mean change score pre to 3 months post: number analyzed (Participants) | 4
  mean change score pre to 3 months post | -25.8 (6.7)

2. Primary Outcome: Dimensions of Anger Reactions (DAR)
Description: The DAR is a 7-item scale measuring the frequency, duration, and behavioral response to anger, and anger-related functional impairment on social relationships, health, and work. It was found to have concurrent and discriminant validity, and to correlate highly with measures of functional impairment, in a large sample of treatment-seeking soldiers who had served in Iraq or Afghanistan. Score range is from 0-56, with higher score reflecting greater problems with anger. Positive change score reflects increase in anger interference from baseline to post-treatment; negative change score reflects decrease in anger interference from baseline to post-treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VETNET
Number analyzed (Participants) | 5
units on a scale
  Baseline | 32 (13.5)
  Post-treatment | 37.8 (12.8)
  3 months post-treatment: number analyzed (Participants) | 4
  3 months post-treatment | 18.3 (10.3)
  mean change score from baseline to post-treatment | 5.8 (5.8)
  mean change score from baseline to 3 months post-treatment: number analyzed (Participants) | 4
  mean change score from baseline to 3 months post-treatment | -9.5 (5.8)

3. Primary Outcome: The Appetitive Aggression Scale (AAS)
Description: This scale has two parts. Part 1 is a 17-item scale that asked participants to mark whether they have engaged in or witness specific violent acts. 15 of these items measure acts that could reflect appetitive aggression (".made another person scream in pain"), and two are more clearly reactive ("...defended yourself in a fight"). If a participant endorses having engaged in any of the 15 potentially appetitive aggressive behaviors, then Part 2 is administered. Data from Part 2 is what is presented here. Part 2 is a 19-item scale that evaluates (yes or no) whether the participant enjoys engaging in violence. Only the first 15 items are scored because these reflect appetitive aggression (the last 4 items evaluate reactive aggression). Total score on Part 2 ranges from 0 to 15, with higher score reflecting greater appetitive aggression. Negative change score reflects decreases in appetitive aggression from baseline to post-treatment; positive change scores reflect increases.
Time Frame: Change in total score from baseline to end of treatment (approximately 10-12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VETNET
Number analyzed (Participants) | 5
units on a scale
  Baseline | 8.6 (3.3)
  post-treatment | 7.8 (3.1)
  mean change score baseline to post-treatment | -0.8 (0.84)

4. Primary Outcome: Beck Depression Inventory (BDI-2)
Description: The BDI-2 is a 21-item scale that evaluates symptoms of depression. Total score range is from 0 to 63, with higher scores indicating greater depression. Negative change scores reflect decrease in depression from pre to post treatment; positive change scores reflect increase in depression from pre to post treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VETNET
Number analyzed (Participants) | 5
units on a scale
  Baseline | 19.2 (5.5)
  post-treatment | 13.2 (7.9)
  3 months post-treatment: number analyzed (Participants) | 4
  3 months post-treatment | 11.3 (8.8)
  mean of change score from baseline to post-treatment | -6 (6.6)
  mean of change score from baseline to 3-months post-treatment: number analyzed (Participants) | 4
  mean of change score from baseline to 3-months post-treatment | -5.8 (9.3)

5. Secondary Outcome: The Moral Injury Events Scale (MIES)
Description: The MIES is an 11-item scale that measures moral injury associated with experiences during military service. Statements related to distress or feelings of betrayal related to potentially morally injurious events are rated on a 6 point scale ranging from 1 (strongly agree) to 6 (strongly disagree). Score range is 11 to 66, with higher scores reflecting greater moral injury. Positive change scores reflect increase in moral injury from pre to post treatment; negative change scores reflect decrease in moral injury from pre to post treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VETNET
Number analyzed (Participants) | 5
units on a scale
  Baseline | 60.4 (16.6)
  post-treatment | 63.6 (25.1)
  3 months post-treatment: number analyzed (Participants) | 4
  3 months post-treatment | 61.3 (14.7)
  mean change score baseline to post-treatment | 3.2 (21.5)
  mean change score baseline to 3 months post-treatment: number analyzed (Participants) | 4
  mean change score baseline to 3 months post-treatment | -4.3 (14.4)

6. Secondary Outcome: Revised Conflict Tactics Scales (CTS2)
Description: The CTS2 includes 78 items measuring the use of psychological and physical attacks by the participant. Participants answer how often these behaviors were perpetrated by them within a specified time period: 0 (never); 1 (once); 2 (twice); 3 (3-5 times); 4 (6-10 times); 5 (11-20 times); 6 (more than 20 times). The original CTS2 instructions will be modified to more appropriately reflect the goals of this study: 1) the target of the behavior will be expanded from "partner" to "anyone"; and 2) the time frame of the response will be reduced from one year to three months to detect potential changes associated with treatment. Two subscale scores were used for these analyses: Psychological Aggression (range = 0 to 48) and Physical Assault (range = 0 to 72), with higher scores reflecting greater use of aggression.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VETNET
Number analyzed (Participants) | 5
units on a scale
  Baseline Psychological Aggression | 8.6 (5.9)
  Post-treatment psychological aggression | 8.6 (7.3)
  3 months post-treatment psychological aggression: number analyzed (Participants) | 4
  3 months post-treatment psychological aggression | 1.8 (2.2)
  mean change score psychological aggression baseline to post-treatment | 0.0 (8.7)
  mean change score psychological aggression baseline to 3 months post-treatment: number analyzed (Participants) | 4
  mean change score psychological aggression baseline to 3 months post-treatment | -6.5 (4.8)
  baseline physical assault | 3.4 (7.1)
  post-treatment physical assault | 2.0 (4.5)
  3 months post-treatment physical assault: number analyzed (Participants) | 4
  3 months post-treatment physical assault | 0.0 (0.0)
  mean change score physical assault baseline to post-treatment | -1.4 (9.3)
  mean change score baseline to 3 months post-treatment: number analyzed (Participants) | 4
  mean change score baseline to 3 months post-treatment | -4.3 (7.8)

7. Secondary Outcome: Trauma-Related Guilt Index (TRGI)
Description: Guided by appraisal theories of emotion, the 32-item TRGI is an index of guilt associated with the experience of trauma. Participants rate statements on a 5-point scale ranging from extremely true/extremely guilty (4) to not at all true/not guilty at all (0). Total scores range from 0 to 128, with higher scores reflecting greater trauma-related guilt.
Time Frame: Change in total score from baseline to end of treatment (approximately 10-12 weeks)
Population: An error was made in administration of the TGRI such that only the first page of a two page measure was given to participants. None of the subscales of the TGRI could be computed with the first page items only. As such, no participant data could be analyzed for this measure.
Arm/Group | VETNET
Number analyzed (Participants) | 0

8. Secondary Outcome: Interpersonal Needs Questionnaire (INQ)
Description: Based upon the Interpersonal Theory of Suicide (Joiner Jr et al., 2009), the INQ measures two proximal causes of the desire for suicide: Thwarted belongingness and Perceived burdensomeness. Participants rate each of the 15 items on a scale of 1 (not at all true for me) to 7 (very true for me). Total scores range from 15 to 105, with greater scores reflecting higher levels of suicide-related cognitions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VETNET
Number analyzed (Participants) | 5
units on a scale
  Baseline | 48.6 (17.7)
  post-treatment | 36.0 (11.2)
  3 months post-treatment: number analyzed (Participants) | 4
  3 months post-treatment | 25.0 (4.2)
  mean change score baseline to post-treatment | -12.6 (14.1)
  mean change score baseline to 3 months post-treatment: number analyzed (Participants) | 4
  mean change score baseline to 3 months post-treatment | -19.3 (15.2)

ADVERSE EVENTS:
Time Frame: 6 months: Veterans completed a baseline assessment, 10-12 weekly sessions of treatment over approximately 2 1/2 to 3 months, a post-treatment assessment, and then completed questionnaires at 3 months post-treatment.
Arm/Group | VETNET
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03777553/Prot_000.pdf
  • Informed Consent Form (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT03777553/ICF_001.pdf